CLINICAL TRIAL: NCT06041386
Title: A Prospective, Real-World, Interventional Study To Evaluate The Effect Of Mepolizumab On Achieving Clinical Remission In Participants With Severe Asthma
Brief Title: REIMAGINE - Real World EvaluatIon of Mepolizumab in Severe Asthma achievinG on Treatment clinIcal remissioN, a prospEctive Study
Acronym: REIMAGINE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 219871
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Severe asthma; Eosinophilic phenotype; Oral corticosteroids (OCS); Asthma exacerbations; Clinical remission; NUCALA; Mepolizumab
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Masking Description: There will be no masking in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Group 1 (Other): Participants with a clinical diagnosis of Severe asthma prescribed Mepolizumab as part of routine care.
  Interventions: Drug: Mepolizumab; Other: Spirometry

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab will be prescribed based on physician decision.
Other: Spirometry — Lung function via spirometry will be collected.

SUMMARY:
This is a prospective, real-world, single arm, global, multi-centre study to evaluate the effect of timely treatment with mepolizumab (NUCALA) to achieve clinical remission in adult participants with severe asthma with an eosinophilic phenotype (SA-EP).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a confirmed asthma diagnosis and has been prescribed NUCALA by their physician for the treatment of asthma, as per local label. NUCALA can be initiated up to 7 days prior to study enrollment.
* No NUCALA use in the 6 months prior to enrollment.
* Participants with greater than or equal to (≥)60 percentage (%) predicted forced expiratory volume in 1 second (FEV1) and less than or equal to (≤)4 exacerbations per year, as confirmed by the physician.
* Other local prescription criteria of NUCALA not described above at NUCALA initiation (e.g., local reimbursement criteria).
* Written informed consent

Exclusion Criteria:

* Investigator concerns about participant's willingness to adhere to biologic treatment for any reason (e.g., cost, behavior, difficulty with access to healthcare)
* Participants currently on maintenance OCS or intramuscular corticosteroids.
* Participants using omalizumab, reslizumab, dupilumab, tezepelumab, or benralizumab within the 6 months prior to enrollment
* Participants participating in an interventional study with a treatment intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2028-06-14 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of Participants Achieving 4-Component Clinical Remission | At month 12
  4-component clinical remission is defined as (a) No clinically significant asthma exacerbations (b) No OCS use for asthma (c) Well controlled asthma based on an Asthma Control Test (ACT) (d) No clinically significant deterioration of lung function.

SECONDARY OUTCOMES:
Annualized Rates of Clinically Significant Asthma Exacerbations (CSE) and CSE Leading to Hospitalization/ Emergency Room (ER) Visits | At month 12
  CSE is defined as a deterioration in asthma requiring (1) the initiation of systemic corticosteroids and/or (2) an ER visit and/or hospital admission.
Percentage of Participants Achieving OCS Sparing Remission | At month 12
  OCS sparing is defined as (a) No clinically significant asthma exacerbations during the period of interest (b) No OCS use for asthma at the time point of interest.
Percentage of Participants Achieving 3-Component Clinical Remission | At month 12
  3-component clinical remission is defined as (a) No clinically significant asthma exacerbations (b) No OCS use for asthma (c) Well controlled asthma based on an ACT
Mean Change from Baseline in Mini-Asthma Quality of Life Questionnaire (AQLQ) Overall Score | Baseline and at month 12
  The mini-AQLQ overall score is a reduced version of the AQLQ which includes 15 items. The minimally clinically important difference (MCID) is 0.5. The response options for each item are on an equidistant scale of 7 points, where 1 corresponds to the maximum disability and 7 to the absence of disability

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (60):
- United States (27):
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Glenn Dale, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Linwood, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Cypress, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, McKinney, Texas
- Belgium (2):
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Liège
- Canada (3):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
- France (6):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
- Germany (6):
  - GSK Investigational Site, Aachen
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Darmstadt
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hohenstein-Ernsttal
  - GSK Investigational Site, Schleswig
- Italy (7):
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Monserrato CA
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Pieve Di Soligo TV
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano
  - GSK Investigational Site, Verona
- Japan (3):
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Tokyo
- Poland (3):
  - GSK Investigational Site, ?Od?
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/